CLINICAL TRIAL: NCT04288141
Title: HERdi PREDICT: A Pilot Study to Measure the Expression of the HER2-HER3 Dimer in Samples From Patients With HER2 Positive Breast Cancer Receiving HER2 Targeted Therapies
Brief Title: A Study to Measure the Expression of the HER2-HER3 Dimer in Tumour and Blood (Exosomes) Samples From Patients With HER2 Positive Breast Cancer Receiving HER2 Targeted Therapies
Acronym: HERdi PREDICT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: HERdi PREDICT
Record Dates: First submitted 2020-02-14; First posted 2020-02-28 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: HER2-positive Breast Cancer
Keywords: FLIM-FRET; HER2-HER3 dimer; Exosomes; Predictive biomarkers
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participant derived tumour samples, exosomes (extracted from serum samples), Peripheral blood mononuclear cells (PBMCs) and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Early HER2 positive breast cancer: Study participants in Group 1 will include patients prescribed neoadjuvant systemic therapy (including trastuzumab and pertuzumab) by their treating oncologist for a diagnosis of HER2 positive early breast cancer.
  Interventions: Other: Acquisition of blood samples and tumour tissue samples (biopsies)
- Group 2: Metastatic HER2 positive breast cancer: Study participants in Group 2 will include patients prescribed systemic therapy (including trastuzumab and pertuzumab) by their treating oncologist for a diagnosis of HER2 positive metastatic breast cancer.
  Interventions: Other: Acquisition of blood samples and tumour tissue samples (biopsies)

INTERVENTIONS:
Other: Acquisition of blood samples and tumour tissue samples (biopsies) — Acquisition of blood samples and tumour tissue samples (biopsies) in a sequential manner as participants proceed through HER2-directed therapy as prescribed by their oncologist.

SUMMARY:
The treatment of breast cancer is determined by its 'receptor (or signal) status'. Receptors are signals present on all cells and if abnormal can drive cancer growth. One of the signals that can drive breast cancer growth is the HER2 receptor/signal. One quarter of all breast cancers are found to have too many HER2 signals i.e. HER2-positive breast cancer.

HER2 is a member of the HER-family which constitutes HER1,HER2,HER3,and HER4 signals. Currently, tests can identify breast cancers with too much HER2, from a biopsy, so a cancer doctor can prescribe anti-HER2 treatment to block these signals. These drugs have improved survival rates in HER2-positive breast cancer. Members of the HER family can also 'pair' with each other to activate signals that encourage cancer growth. For example, HER3 naturally 'pairs' with HER2. Though anti-cancer drugs have been developed to target this pairing, the current method of patient selection is not developed to detect pairing of signals in tissue biopsies. A specialist imaging technique called FLIM-FRET (FLIM- Fluorescence Lifetime Imaging Microscopy; FRET- Forster resonance energy transfer) can identify signal pairing on cancer cells from tissue, and potentially, from blood samples.

This study involves having blood tests while participants receive anti-HER2 treatment. The investigators will also seek permission to take samples of cancer tissue from the biopsies that were already carried out, e.g. at diagnosis. Some participants may need an additional biopsy, which will be discussed with participants prior to consent. This study will use the specialist FLIM-FRET technique to measure the signal pairing in tumour samples and blood samples. Investigators will measure if the levels of signal pairing from blood are the same as that from tissue, which could lead to bloods tests being used to select patients for anti-HER2 treatments, instead of invasive tissue biopsies. Changes in signal pairing may also help to predict if a cancer is becoming resistant to treatment.

DETAILED DESCRIPTION:
The study will recruit 40 participants to two groups as outlined below:

Group 1: Early HER2 positive breast cancer (20 patients) Group 2: Metastatic HER2 positive breast cancer (20 patients)

The two groups represent the natural spectrum of breast cancer in its clinical presentation.

GROUP 1: EARLY BREAST CANCER

Group 1 will include patients with early HER2 positive breast cancer recommended to receive neo-adjuvant chemotherapy inclusive of HER2 directed therapy (trastuzumab + pertuzumab), prior to proceeding to curative surgery. All participants are expected to have had a diagnostic core biopsy and definitive breast surgery on completion of neoadjuvant chemotherapy as standard of care. Blood samples will be obtained for biomarker analysis in exosomes. Participants in Group 1 A will be requested to have a biopsy on completion of anthracycline based chemotherapy and prior to commencing on HER2-directed therapy.

Group 1 A: Participants in Group 1 commencing treatment with anthracycline based chemotherapy for up to 4 cycles followed by a switch in treatment to taxane based chemotherapy in combination with HER2 directed therapy (trastuzumab + pertuzumab) for up to 4 cycles

Group 1 B: Participants in Group 1 commencing treatment with taxane based systemic therapy in combination with HER2 directed therapy (trastuzumab + pertuzumab) for up to 6 cycles:

GROUP 2: METASTATIC BREAST CANCER:

Group 2 will include patients will include participants recommended commencing any line of palliative systemic therapy inclusive of a HER2 directed therapy by their treating oncologist. All participants are expected to have had a diagnostic core biopsy. Blood samples will be obtained for biomarker analysis in exosomes.

ELIGIBILITY:
Inclusion Criteria:

1. Female or Male aged 18 years or above.
2. Histologically documented breast cancer. In participants with metastatic breast cancer (Group 2), the biopsy should have been obtained following or at the time of diagnosis of metastatic breast cancer. (refer to inclusion criteria 10 for group 2 specific criteria)
3. HER2 positive breast cancer, to be established by immunohistochemistry and confirmed by fluorescence in situ hybridisation or dual in situ hybridisation in borderline cases as per standard of care guidelines.
4. Confirmation of availability of sufficient tumour tissue (from diagnostic core biopsy) for biomarker analysis (Refer to study laboratory manual)
5. Fit for treatment with chemotherapy in combination with HER2 targeted therapy as per investigator discretion
6. Life expectancy of 12 weeks or more.
7. Participant is willing and able to give informed consent for participation in the study and in the investigator's opinion, is able and willing to comply with all study requirements.
8. Participant willing to undergo additional biopsies when required i.e. Group 1A and Group 2
9. Willing to allow his or her general practitioner to be notified of participation in the study [optional].
10. Group 2 specific criteria

    1. The pre-treatment tumour sample for biomarker analysis in group 2 will be acquired from the diagnostic biopsy acquired when participants were first diagnosed with metastatic HER2 positive breast cancer. The biopsy should have been acquired following or at the time of the diagnosis of metastatic breast cancer (i.e. cannot use tumour tissue acquired during a prior diagnosis of early/locally advanced breast cancer for this study's biomarker analysis). The biopsy may be acquired from a breast mass or a metastatic site. If a biopsy following or at the time of the diagnosis of metastatic breast cancer has not been carried out, a study specific biopsy will need to be organised.
    2. Only patients recommended first line treatment with a taxane, trastuzumab and pertuzumab by their physician, are eligible. Potential participants being considered for treatment with any other treatment combinations with HER2 targeted therapies will not be considered eligible.

Exclusion Criteria

1. Significant thrombocytopaenia or abnormal clotting screen or any other condition that would contraindicate a tissue biopsy if this were required, in the investigator's opinion.
2. Participant unwilling to undergo study required tissue biopsies and blood sampling.
3. Any other significant underlying condition or comorbidity which, in the opinion of the investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study or the participant's ability to participate in the study.
4. Inability of participant to co-operate with study procedures as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: Early HER2 positive breast cancer and prescribed neoadjuvant chemotherapy including trastuzumab and pertuzumab as per physician discretion.
  Group 2: Metastatic HER2 positive breast cancer and prescribed chemotherapy including trastuzumab and pertuzumab as per physician discretion.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Compare HER2-HER3 dimer expression as detected by FLIM-FRET (% positive for HER2-HER3 dimer expression with FRET efficiency ≥8.56%) to HER2 over-expression (% positive for HER2 over-expression by IHC ± FISH) in patient-derived tumour samples. | Group 1: Baseline biopsy and definitive surgical specimen. Group 2: Baseline biopsy.

SECONDARY OUTCOMES:
Describe the range of FRET efficiency determined by measuring tumoural HER2-HER3 dimerisation as a continuous variable. | Group 1: Baseline biopsy and definitive surgical specimen. Group 2: Baseline biopsy.
Compare the HER2-HER3 dimer expression level in tumour samples to matched blood samples (exosomal expression) as detected by FLIM-FRET. | Each cycle (C) is 21 days (D). Group 1A & Group 1B: Baseline biopsy,definitive surgical specimen and paired blood samples. Group 1A: Also in matched interim tumour and blood sample (C4 D14-21). Group 2: Baseline biopsy and blood sample
Compare HER2 expression in blood samples (exosomes) by protein detection assays e.g. dot blots to HER2 status in matched tumour tissue as determined by IHC ± FISH. | Each cycle (C) is 21 days (D). In group1 HER2 expression in matched participant tumour tissue and blood will be compared at baseline and immediately after completion of neoadjuvant therapy/surgery. In Group 2, to be assessed at baseline only.
Determine the range of measurable exosomal FRET efficiency determined by measuring exosomal HER2-HER3 dimer expression. | Each cycle (C) is 21 days (D). In group1a: Baseline, C2 D1, C5 D1, C6 D1 and C8 D21-42. In Group 1b: Baseline, C2 D1, C6 D21-42, Group 2: Baseline, C2 D1, C4/5 D1.
Determine if patient derived tumour and blood samples (exosomes) demonstrate a change in HER2-HER3 dimer expression in response to systemic HER2-directed therapy (% positive for change in HER2-HER3 dimer expression). | Each cycle (C) is 21 days (D). In group1a: Baseline, C2 D1, C5 D1, C6 D1 and C8 D21-42. In Group 1b: Baseline, C2 D1, C6 D21-42, Group 2: Baseline, C2 D1, C4/5 D1. In tumour at baseline, C4 D14-21 (group 1a only) & immediately after surgery(group 1 only)
Determine the statistical association of FRET efficiency (at baseline and any subsequent changes) determined by measuring tumoural HER2-HER3 dimer expression with radiological and pathological responses to systemic treatment. | Each cycle (C) is 21 days (D). HER2-HER3 dimer measured in tumour at baseline, C4 D14-21 (group 1a only) & immediately after surgery (group 1 only). Radiology imaging as standard of care (SoC) during course of the study.
Determine the statistical association of FRET efficiency (at baseline and any subsequent changes) determined by measuring exosomal HER2-HER3 dimer expression with radiological and pathological responses to systemic treatment | Each cycle (C) is 21 days (D). In group1a: Baseline, C2 D1, C5 D1, C6 D1 and C8 D21-42. In Group 1b: Baseline, C2 D1, C6 D21-42, Group 2: Baseline, C2 D1, C4/5 D1. Pathological response immediately after surgery(group 1 only). Radiology imaging as SoC
Determine the statistical association of the levels of expression of immune cell markers (at baseline and any subsequent changes) with radiological and pathological responses to systemic treatment. (OPTIONAL CONSENT-Guy's hospital site only). | Each cycle (C) is 21 days (D). In group1a: Baseline, C2 D1, C5 D1, C6 D1 and C8 D21-42. In Group 1b: Baseline, C2 D1, C6 D21-42, Group 2: Baseline, C2 D1, C4/5 D1. Pathological response immediately after surgery(group 1 only). Radiology imaging as SoC.
Determine feasibility of using exosomal expression testing in a National Health Service (NHS) practice. | On study completion
  1. Determine the percentage of participant derived blood samples processed appropriately in the clinical setting and transported to the central laboratory for exosome analysis.
  2. Describe the reasons for obtaining unsuitable participant derived blood samples from clinics.
  3. Determine the percentage of participant derived blood samples that are successfully analysed for biomarker expression i.e. % of blood samples demonstrating exosomal isolation, % of blood samples demonstrating HER2-HER3 dimerisation.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Guy's Cancer Centre, Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No